CLINICAL TRIAL: NCT03789305
Title: Differences in Frail and Non-frail Critically-ill Patients in Functional Outcomes
Acronym: DEFAULT
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Stefan Schaller, Principal Investigator, Technical University of Munich
Other Study IDs: DEFAULT
Record Dates: First submitted 2018-12-25; First posted 2018-12-28 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Critical Care; Rehabilitation; Outcome Assessment; Critical Illness; Frailty; Physical and Rehabilitation Medicine; Exercise Therapy; Intensive Care Unit
Keywords: Early Mobilization; Early Rehabilitation; Functional Status; Functional Outcome; Patient Outcome; Intensive Care; Critical Care Outcomes
MeSH Terms: conditions — Critical Illness; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Critically ill patients admitted to intensive care for more than 48 hours

SUMMARY:
This is a prospective analysis of patient registry data of intensive care patients. The aim is to investigate if frailty is a predictor of decline of functional status of critically ill patients during their hospital stay.

DETAILED DESCRIPTION:
Elderly critical-ill patients with a high frailty level are becoming increasingly important in the ICU and the health system. Especially, questions about the course of the individual proceeding, withhold of therapy and level of care are controversial among caretakers, as outcome and functional independence remain still unclear in these patients.

This applies particularly in view of the fact that large studies such as VIP1 showed an inverse association of high frailty classes with short-term survival.

Our main objective in this study was to focus on functional outcome and independency measured by Barthel Index after ICU stay regarding frailty, the effect of critical care and severity and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* intensive care stay > 48 hours

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to two intensive care units at a university hospital from the Department of Anesthesiology and Intensive Care in Munich, Germany.
Sampling Method: Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Probability not to deteriorate in functional status during the hospital stay | a median of 30 days
  Analysis of the course of functional status measured by the Barthel Score sub-components transfer and ambulation during the hospital stay. The Scale ranges from 0 (no transfer) to 15 (transfer to chair and back) for transfer and from 0 (no ambulation) to 15 (coming into stand and walk 50m without supervision) for ambulation.

SECONDARY OUTCOMES:
Change in Functional status before hospital admission to ICU discharge | a median of 20 days
  Analysis of the change of functional status measured by the Barthel Score sub-components transfer and ambulation from before hospital admission to ICU discharge. The Scale ranges from 0 (no transfer) to 15 (transfer to chair and back) for transfer and from 0 (no ambulation) to 15 (coming into stand and walk 50m without supervision) for ambulation.
Change in Functional status before hospital admission to hospital discharge | a median of 30 days
  Analysis of the change of functional status measured by the Barthel Score sub-components transfer and ambulation from before hospital admission to hospital discharge. The Scale ranges from 0 (no transfer) to 15 (transfer to chair and back) for transfer and from 0 (no ambulation) to 15 (coming into stand and walk 50m without supervision) for ambulation.
ICU length of stay | a median of 11 days
  Duration of stay on intensive care
Hospital length of stay | a median of 30 days
  Duration of stay in the hospital
Rate of discharge disposition to home | 1 day
  Rate of participants being discharged home after the hospital stay.
ICU mortality | a median of 11 days
  Expired during the intensive care stay
Hospital mortality | a median of 22 days
  Expired during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, MHBA, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, School of Medicine, Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be made available to other researchers on reasonable request. A data share agreement will have to be signed by both parties.
  Examples of reasonable requests are:
  * a metaanalysis in the field
  * a research collaboration
  * rerun the analysis Data will only be provided for the purpose requested and may not be used otherwise without authorization/agreement.

REFERENCES:
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Flaatten H, De Lange DW, Morandi A, Andersen FH, Artigas A, Bertolini G, Boumendil A, Cecconi M, Christensen S, Faraldi L, Fjolner J, Jung C, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zaferidis T, Guidet B; VIP1 study group. The impact of frailty on ICU and 30-day mortality and the level of care in very elderly patients (>/= 80 years). Intensive Care Med. 2017 Dec;43(12):1820-1828. doi: 10.1007/s00134-017-4940-8. Epub 2017 Sep 21. PMID 28936626
- [Background] Latronico N, Herridge M, Hopkins RO, Angus D, Hart N, Hermans G, Iwashyna T, Arabi Y, Citerio G, Ely EW, Hall J, Mehta S, Puntillo K, Van den Hoeven J, Wunsch H, Cook D, Dos Santos C, Rubenfeld G, Vincent JL, Van den Berghe G, Azoulay E, Needham DM. The ICM research agenda on intensive care unit-acquired weakness. Intensive Care Med. 2017 Sep;43(9):1270-1281. doi: 10.1007/s00134-017-4757-5. Epub 2017 Mar 13. PMID 28289812